CLINICAL TRIAL: NCT05498402
Title: Effect of Intermediate Airway Management Using an I-gel® on Ventilation Parameters in Simulated Pediatric Out-of-Hospital Cardiac Arrest: Protocol for a Randomized Crossover Trial
Brief Title: Effect of IAM With an I-gel® on Ventilation Parameters in Simulated Pediatric OHCA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Geneve TEAM Ambulances (Other)
Collaborators: ESAMB - College of Higher Education in Ambulance Care (Unknown); Ambulances de la Ville de Sion (Unknown); University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Stuby Loric, Principal Investigator, Geneve TEAM Ambulances
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CPR-6
Record Dates: First submitted 2022-08-09; First posted 2022-08-12 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Pediatric ALL; Cardiac Arrest; Cardiopulmonary Arrest; Resuscitation; Pediatric Emergency Medicine
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Heart Arrest

STUDY DESIGN:
Intervention Model Description: Prospective, multicenter, crossover, simulation-based, randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: Data extraction will be fully automated and the statistician will not know the identity of the participants or the sequence they were allocated to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bag-valve-mask ventilation (Active Comparator): Providers will perform a cardiopulmonary resuscitation, and deliver ventilations using a bag-valve-mask
  Interventions: Device: bag-valve-mask ventilation
- Supraglottic airway device ventilation (Experimental): Providers will perform a cardiopulmonary resuscitation, and deliver ventilations using an i-gel® supraglottic airway device
  Interventions: Device: i-gel ® device

INTERVENTIONS:
Device: i-gel ® device — Ventilations will be delivered through an i-gel ® device
  Arms: Supraglottic airway device ventilation
Device: bag-valve-mask ventilation — Ventilations will be delivered using a bag-valve-mask
  Arms: Bag-valve-mask ventilation

SUMMARY:
Pediatric cardiac arrest occurs most in the prehospital setting. Most of them are due to respiratory failure (e.g., trauma, drowning, respiratory distress), where hypoxia leads to cardiac arrest. Generally, emergency medical services (EMS) first use basic airway management techniques i.e., the use of a bag-valve-mask (BVM) device, to restore oxygenation in pediatric OHCA victims. However, these devices present many drawbacks and limitations. Intermediate airway management, i.e., the use of SGA devices, especially the i-gel® has several advantages. It has been shown to enhance both circulatory and ventilatory parameters. There is increasing evidence that IAM devices can safely be used in children. In two pediatric studies of OHCA, American paramedics had significantly higher success rates with SGA devices than with TI. A neonatal animal model showed that the use of SGA was feasible and non-inferior to TI in this population. However, data regarding the effect of IAM with an i-gel® versus the use of a BVM on ventilation parameters during pediatric OHCA is missing. The hypothesis underlying this study is that, in case of pediatric OHCA, early insertion of an i-gel® device without prior BVM ventilation should improve ventilation parameters in comparison with the standard approach consisting in BVM ventilations.

DETAILED DESCRIPTION:
Pediatric cardiac arrest is a high-risk, low-frequency event associated with death or severe neurological sequelae in survivors. Most occur in the prehospital setting. Despite advances in resuscitation science and survival improvement over the last decades, survival remains low, with only approximately 6% to 20% of children surviving to hospital discharge after pediatric out-of-hospital cardiac arrest (OHCA). Most triggers of pediatric OHCA are respiratory in nature, with sudden infant death syndrome, trauma and drowning among the main etiologies, where hypoxia leads to cardiac arrest. Prompt and effective airway management is therefore paramount when responding to a pediatric OHCA. Any delay in intermediate or advanced airway management has been associated with a decreased chance of survival. The debate about the optimal airway management strategy that should be used in pediatric OHCA is, however, still ongoing.

Generally, emergency medical services (EMS) first use basic airway management techniques i.e., the use of a bag-valve-mask (BVM) device, to restore oxygenation in pediatric OHCA victims. However, these devices present many drawbacks and limitations. First, airtightness must be ensured to enable adequate oxygenation. Second, the use of BVM is associated with gastric air insufflation. This can alter oxygenation by restricting total lung capacity and, consequently, lung compliance. Since decreased lung compliance requires the use of higher pressures to reach the same tidal volume, gastric inflation can indirectly impair venous return. In addition, chest compressions during cardiopulmonary resuscitation (CPR) must be interrupted to provide ventilations when basic airway management devices are used. However, these interruptions decrease coronary and cerebral blood flow and should be minimized as they have been associated with decreased survival both in animals and humans.

On the other hand, advanced airway management, i.e., tracheal intubation (TI), provides optimal airtightness -thereby avoiding gastric inflation and risk of regurgitation- while allowing the provision of asynchronous ventilations during CPR. However, advanced airway management requires advanced skills that must be maintained through regular practice. Depending on the regional context, skilled prehospital providers may not be immediately available, if at all. This is particularly important when taking care of critically ill children, whom many consider difficult to intubate. The failure rate of TI at first attempt in case of pediatric CPR is high, even in the hospital setting, and associated with unfavorable neurological and survival outcomes. Recently, a registry-based study reported these outcomes to be worse after pediatric OHCA when emergency physicians used TI rather than supraglottic airway (SGA) devices. The interpretation of these results is however limited by the lack of data regarding physician experience and TI attempts.

In line with the above listed limitations of basic or advanced airway management devices, intermediate airway management (IAM) i.e., the use of SGA devices [18], could represent a valuable alternative in prehospital settings. One of the best studied SGA devices is the i-gel®, which is both easy and fast to insert, and provides high leak pressures. Its use is associated with a high overall success rate and is easily remembered. Regurgitation and aspiration are not more frequent with IAM devices than with TI and are much less likely than when a BVM device is used. The use of an i-gel® enables continuous chest compressions in most cases, and a higher first rate of successful initial ventilation. This device has been found to increase the chest compression fraction (CCF) and improve ventilations parameters in an adult model of OHCA. In real OHCA, compared to TI, similar outcomes at 30 days and 6 months were found.

There is increasing evidence that IAM devices can safely be used in children. In two pediatric studies of OHCA, American paramedics had significantly higher success rates with SGA devices than with TI. A neonatal animal model showed that the use of SGA was feasible and non-inferior to TI in this population. However, data regarding the effect of IAM with an i-gel® versus the use of a BVM on ventilation parameters during pediatric OHCA is missing. The hypothesis underlying this study is that, in case of pediatric OHCA, early insertion of an i-gel® device without prior BVM ventilation should improve ventilation parameters in comparison with the standard approach consisting in BVM ventilations.

For this purpose, a prospective, multicenter, crossover, randomized controlled trial with two groups will be conduct in four EMS in different French-speaking part of Switzerland. This will be a simulation-based study.

ELIGIBILITY:
Inclusion Criteria:

* Being a registered EMT, or paramedic

Exclusion Criteria:

* Member of the study team

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2023-01-30 (Actual); Primary Completion 2023-06-13 (Actual); Study Completion 2023-06-13 (Actual)

PRIMARY OUTCOMES:
Alveolar ventilation per minute | 10 minutes of scenario
  It will be determined by subtracting the dead space volume from each ventilation, then multiplied by the ventilations' count, and divided by the duration of the ventilation period (i.e., 10 minutes - time to the first ventilation). The simulated child's dead space volume corresponds to about 27 ml using the formula proposed by Numa and Newth. The physiological tidal volume range is of 5 to 8 ml/kg, corresponding to 45 to 72 ml for the simulated child's.

SECONDARY OUTCOMES:
The proportion, and number of ventilations below, within and over the target volume | 10 minutes of scenario
  The target volume is 45 to 72 ml.
The time to the first efficient ventilation | 10 minutes of scenario
  Corresponds to the time elapsed between T0 (the first therapeutical action) and the first efficient ventilation (equal or superior to 45 ml)
The time to the first compression | 10 minutes of scenario
  Corresponds to the time elapsed between T0 (the first therapeutical action) and the first compression
The chest compression fraction | 10 minutes of scenario
  Corresponds to the time during which compressions have been performed on the total CPR time
The chest compression rate | 10 minutes of scenario
  Corresponds to the number of compressions delivered by minute
The proportion of chest compressions below, within and over the target rate | 10 minutes of scenario
  The target rate is 100 to 120 compressions per minute
The compression depth | 10 minutes of scenario
  Corresponds to the depth of the chest compressions
The proportion of chest compressions below and within the target depth | 10 minutes of scenario
  The threshold is 4.3 cm (corresponding to one third of the manikin's measured anteroposterior chest depth)
The proportion of complete chest recoil | 10 minutes of scenario
  Corresponds to the proportions of compression released to at least 5 mm from the baseline
The time to first epinephrine injection | 10 minutes of scenario
  Corresponds to the time elapsed between the first therapeutical action (T0) and the time-point where epinephrine is administered
The proportion of scenarios in which epinephrine is administered within 5 minutes | 10 minutes of scenario
  The part of scenarios where epinephrine was administered following the recommandations

CONTACTS AND LOCATIONS:
Overall Officials: Loric Stuby, Principal Investigator — Genève TEAM Ambulances
Locations (4):
- Switzerland (4):
  - ACE Genève Ambulances, Chêne-Bougeries, Canton of Geneva
  - Ambulances de la Ville de Sion, Sion, Valais
  - Genève TEAM Ambulances, Geneva
  - SK Ambulances, Geneva

IPD SHARING:
Plan to Share IPD: Yes
The study protocol will be published in a peer-reviewed journal. The data will be freely available on Yareta
Supporting Information: Study Protocol
Time Frame: We plan to submit the protocol for publication in the second semester of 2022. The study's data will be accessible once the results submitted for publication
Access Criteria: The data would be accessible freely on Yareta

REFERENCES:
- [Derived] Stuby L, Bourgeois L, Tinembart JM, Muhlemann E, Thurre D, Siebert JN, Suppan L. Effect of intermediate airway management on ventilation parameters in simulated paediatric out-of-hospital cardiac arrest: a multicentre randomised crossover trial. Swiss Med Wkly. 2025 May 16;155:4079. doi: 10.57187/s.4079. PMID 40450752
- See also: Whole project website — https://swiss-cpr-studies.ch/